CLINICAL TRIAL: NCT03555214
Title: Efficacy of Manual Therapy for the Treatment of Chronic Migraine.
Brief Title: Efficacy of Manual Therapy for the Treatment of Migraine.
Acronym: MT-Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ID0024
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Migraine
Keywords: migraine; manual therapy
MeSH Terms: conditions — Migraine Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Manual Therapy based on soft tissue (Experimental)
  Interventions: Other: Manual Therapy based on soft tissues
- Control Group (Placebo Comparator)
  Interventions: Other: Control group
- Manual Therapy based on structural techniques (Experimental)
  Interventions: Other: Manual Therapy based on structural techniques
- Manual Therapy based on soft tissue and structural techniques (Experimental)
  Interventions: Other: Manual Therapy based on soft tissues and structural techniques

INTERVENTIONS:
Other: Manual Therapy based on soft tissues — Manual Therapy:
  1. Technique of suboccipital inhibition.
  2. Cranial frontal technique.
  3. Cranial sphenoid technique.
  4. Cranial fourth ventricle technique.
  5. Antero-posterior abdominal-sacral technique.
  Arms: Manual Therapy based on soft tissue
Other: Control group — Placebo treatment:
  The patient remains supine and the therapist sits on a stool at the bedside with the forearms resting on the couch. Both hands are placed on the posterolateral part of the patient's head and the position is maintained for 10 minutes without exerting any force or movement.
  Arms: Control Group
Other: Manual Therapy based on structural techniques — Manual Therapy:
  1. Technique of manipulation of the occipito-atlanto-axoidea joint (OAA).
  2. Articulation technique of the high cervical spine (C0-C1).
  3. Postero-anterior articular technique of C2-C7 in supine position.
  4. Postero-anterior articular technique of C2-C7 in prone position.
  5. Manipulative technique of the flapper C7-T1.
  6. Dorsal spinal manipulative technique (T1-T8).
  7. Lumbosacral global manipulative technique.
  Arms: Manual Therapy based on structural techniques
Other: Manual Therapy based on soft tissues and structural techniques — Manual Therapy:
  1. Technique of suboccipital inhibition.
  2. Cranial frontal technique.
  3. Cranial sphenoid technique.
  4. Cranial fourth ventricle technique.
  5. Antero-posterior abdominal-sacral technique.
  6. Technique of manipulation of the occipito-atlanto-axoidea joint (OAA).
  7. Articulation technique of the high cervical spine (C0-C1).
  8. Postero-anterior articular technique of C2-C7 in supine position.
  9. Postero-anterior articular technique of C2-C7 in prone position.
  10. Manipulative technique of the flapper C7-T1.
  11. Dorsal spinal manipulative technique (T1-T8).
  12. Lumbosacral global manipulative technique.
  Arms: Manual Therapy based on soft tissue and structural techniques

SUMMARY:
Introduction According to the World Health Organization (WHO) at least 47% of adults have suffered from headache in the last year. The headache is not only painful but also disabling, it can be accompanied by social and personal problems, with a decrease in the quality of life and with economic losses. Migraine affects a large number of people and, if the predisposing factors are not controlled, it can become chronic. Once the chronification point of migraine has arrived, it seriously affects the quality of life of people, both in the workplace, social and leisure.

objective Perform the application of a manual therapy treatment based on protocols that include techniques already proven to improve different areas of impact in patients with migraine. To evaluate various aspects, we will include the intensity of pain, the frequency of episodes, anxiety and depression, quality of life, etc ... and the limitations or disability that it produces.

Material and methods This is a prospective, single-blind, randomized study with patients diagnosed with migraine. The sample will be distributed in 4 groups: a) experimental group that will receive combined treatment of soft tissues with techniques evidenced independently; b) Group that will receive independent structural techniques; c) the group that will receive the set of protocols a and b; d) and the placebo control group.

Evaluation An initial assessment will be carried out, another at the end of the treatment and another follow-up one month after the end of the treatment. In addition, the evaluation will include the following instruments: the HDI scale (Headache Disability Inventory), the MIDAS scale (Migraine Disability Assessment Scale), the SF-36 Questionnaire, the EVA Scale (Visual-Analogue Scale), the HIT-6 Questionnaire, the BDI Questionnaire (Beck Inventory Depression), the STAI Questionnaire (The State-Trait Anxiety Inventory), the change perceived after the treatment and medication intake.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 4 migrainous crises per month, following the criteria established by the IHS
* history of episodes of more than a year of evolution
* use of stable medication during the four weeks prior to the start of the study
* between 18 and 60 years old

Exclusion Criteria:

* currently being in physiotherapy preventive treatment
* being in the process of pharmacological adaptation
* have artery-vertebral involvement problems (bone degeneration, metabolic or musculoskeletal problems that involve vertebral artery risk)
* suffer from dizziness
* suffering dizziness or unbalanced tension.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Intensity of Pain | 8 weeks
  Visual Analog Scale. It is a commonly used and validated instrument in the interpretation of pain intensity. In a line of 10 cm, divided by numbers from 0 to 10, the patient marks the intensity of the pain, being 0 "absence of pain" and 10 "worst pain imaginable".

SECONDARY OUTCOMES:
Disability | 8 weeks
  Headache Disability Inventory (HDI). Questionnaire developed by G.P. Jacobson et al. to quantify the impact of disability due to headache in daily life. The objective is to identify the difficulties that the patient experiences due to headaches. It consists of two questions: 1) intensity of pain (mild, moderate and severe), and 2) frequency (once a month, more than 1 and less than 4 times a month, and once a week). In addition, it includes 25 items with two subscales, one emotional (13 items) and another functional (12 items) with three possible answers ("no" 0 points, "sometimes" 2 points, "yes" 4 points). The maximum score is 100 points, with 0 "no disability" and 100 "maximum disability".
Health status | 8 weeks
  SF-36. It consists of 36 items with the following scales: Physical function (items 3a, 3b, 3c, 3d, 3e, 3f, 3g, 3h, 3i, 3j), Physical role (items 4a, 4b, 4c, 4d), Corporal pain ( items 7, 8), General Health (items 1, 11a, 11b, 11c, 11d), Vitality (items 9a, 9e, 9g, 9i), Social function (items 6, 10), Emotional role (items 5a, 5b, 5c) and Mental Health (items 9b, 9c, 9d, 9f, 9h). Includes an item on the change in the general health status with respect to the previous year (item 2). To calculate the score, we must first homogenize the address of the answers by re-coding the items that require it, so that "the higher the score, the better the health condition", then the calculation of the sum of the items of each scale and, finally, the linear transformation of raw scores on a scale of 0 (worst health status for that dimension) to 100 (the best health status).
Headache Impact | 8 weeks
  Headache Impact Test-6 (HIT-6). Published by Ware et al. To measure the impact of headache. The score is calculated as follows: never (6 points), few times (8 points), sometimes (10 points), very often (11 points) and always (13 points). With a total of 49 or less points is considered "little or no impact", between 50-55 "some impact", between 56-59 "significant impact" and 60 or more "very severe impact".
Depression | 8 weeks
  Beck Inventory Depression. It is a questionnaire used to measure the severity of depression in adolescents and adults. Published by Beck et al. And reviewed in 1996,1 questions that include a cognitive-affective factor and a somatic-motivational factor, collecting symptoms such as hopelessness, irritability, dissatisfaction with oneself, changes in the sleep pattern, loss of energy, difficulty of concentration and fatigue-fatigue. In 1972, Beck et al. they developed the short form with 13 items. Each item is valued from 0 to 3, with a total score of 39. The cut-off points recommended by the American Psychiatric Association are: 0-4 absent or minimal, 5-7 mild, 8-15 moderate,> 15 severe.
Change perceived after treatment | 8 weeks
  Global Impression Change Scale. To assess the change perceived after the treatment, patients are asked to rate their perception of change in the Global Impression Change Scale of the patient, and a questionnaire with a question and 7 alternatives, being 1 "maximum change" and 7 "Nothing of change".
Anxiety | 8 weeks
  State-Trait Anxiety Inventory (STAI). Questionnaire developed by Spielberger et al.1 showed that it is the seventh most used questionnaire in Spain.
  It consists of 40 items and they are valued on Likert scales of four points. It is divided into two sections: anxiety-state (items 1 to 20) and anxiety-trait (items 21 to 40); the first in relation to an emotional state that can vary in intensity over time, and the second, measures the tendency to anxiety and to perceive situations as threatening. As a result, a score <30 indicates a low level of anxiety, between 30 and 44 points, average anxiety level, and> 44 points, high anxiety level.
Medication intake | 8 weeks
  All patients were asked about medication intake
Migraine Disability | 8 weeks
  Disability caused by migraine was assessed using the Migraine Disability Assessment (MIDAS). On the one hand, it is composed of five questions about lost or less productive days in relation to paid work (questions 1 and 2), housework (questions 3 and 4) and family, social or recreational activities (question 5) due to headaches. The total score is the sum of the days of the 5 questions. On the other hand, it contains 2 clinically relevant questions about headache frequency and pain intensity, . Finally, the score is divided into grade I = 0-5 points, grade II = 6-10 points, grade III = 11-20 points, and grade IV = 21 or more points. In this way, disability is divided into grade I (slight limitations and few treatment needs in patients), grade II (moderate limitations and moderate treatment needs and grades III and IV (serious limitations and great treatment needs).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy, Valencia, Spain